CLINICAL TRIAL: NCT01483716
Title: A Trial of Rehabilitation in Obesity Hypoventilation Syndrome (OHS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Swapna Mandal, Clinical Research Fellow, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/LO/1481
Record Dates: First submitted 2011-11-30; First posted 2011-12-01 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Obesity Hypoventilation Syndrome
MeSH Terms: conditions — Obesity Hypoventilation Syndrome | interventions — Rehabilitation

ARMS (2):
- Control (No Intervention): NIV alone
- Intervention (Experimental): Rehabilitation arm
  Interventions: Behavioral: Rehabilitation

INTERVENTIONS:
Behavioral: Rehabilitation
  Arms: Intervention

SUMMARY:
Obesity is an escalating problem in the UK and a proportion of these patients have a condition known as Obesity Hypoventilation Syndrome (OHS). This syndrome is associated with symptoms of breathlessness, reduction in exercise capacity, fatigue and headaches. Previous research has shown that patients with this condition tend to use healthcare services more frequently and are often at risk of other diseases such as diabetes mellitus and high blood pressure. Currently, the mainstay of treatment is noninvasive ventilation (NIV), this is a mask ventilator that patients use overnight to improve oxygen levels and remove carbon dioxide (the waste gas of breathing), however this does not fully treat the underlying problem. The research group has shown that NIV helps improve activity and contributes to weight loss in this group of patients. The aim of this research will be to investigate the effect of an exercise and nutrition programme in addition to NIV on weight loss and activity levels compared to NIV alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OHS
* Age >18
* BMI > 30 kg/m2
* Chronic hypercapnia , daytime PaCO2 >6kPa
* FEV1/FVC ≥70%
* Evidence of sleep disordered breathing on overnight studies
* Tolerated NIV > 4hrs on 1st night during initiation of NIV

Exclusion Criteria:

* Hypercapnic respiratory failure secondary to an identifiable cause other than OHS.
* Age <18
* Respiratory acidosis (pH <7.35)
* Wheelchair/bedbound patients
* Cognitive impairment which would prevent the subject from complying with trial protocol
* Unstable coronary artery syndrome
* Patients postintubation or decannulation following treatment requiring acute hypercapnic respiratory failure
* Patients undergoing renal replacement therapy
* Critical peripheral vascular disease
* Disabling locomotor disability preventing participation in exercises involved in the rehabilitation programme
* Pregnancy
* Bariatric surgery planned within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
% Weight loss | 12 months

SECONDARY OUTCOMES:
6 minute walk test | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hart, Study Director — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Mandal S, Suh ES, Harding R, Vaughan-France A, Ramsay M, Connolly B, Bear DE, MacLaughlin H, Greenwood SA, Polkey MI, Elliott M, Chen T, Douiri A, Moxham J, Murphy PB, Hart N. Nutrition and Exercise Rehabilitation in Obesity hypoventilation syndrome (NERO): a pilot randomised controlled trial. Thorax. 2018 Jan;73(1):62-69. doi: 10.1136/thoraxjnl-2016-209826. Epub 2017 Sep 29. PMID 28971973